CLINICAL TRIAL: NCT04319744
Title: The Effectiveness of Video Game Playing Habit in Gaining Video Stylet-mediated Intubation Skill
Brief Title: The Effect of Playing Video Game on Intubation Skill
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Özlem Sezen, Anesthesiology and Reanimation specialist, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: OSezen
Record Dates: First submitted 2020-03-08; First posted 2020-03-24 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Intubation; Airway Management
Keywords: video stylet; airway; video game

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Assistants who have a habit of playing video: Group I:Anesthesia assistants who have a habit of playing video games before Video game will be played for 5 days a day with 0.5 hours mobile phone (Pubg mobile) for those who have previous game experience.
  Intubation training will be provided with video style.Within the scope of this training, 1-All participants will watch videos about Video style application.
  2-Verbal explanation will be made by the responsible and investigators of the study 3- All participants will practice on the model first
  4-Responsible investigators will practice and show on the real patient.
  5-Then all participants will perform the application on the real patient under the supervision of responsible and investigators.
  Tracheal intubation time, success rate, number of interventions will be recorded by responsible and investigators.
  Interventions: Other: other
- Assistants who do not have the habit of playing video: Group II:Anesthesia assistants who do not have the habit of playing video games No video game will be played before intubation with video style for this group.
  Intubation training will be provided with video style. Within the scope of this training, 1-All participants will watch videos about Video style application.
  2-Verbal explanation will be made by the responsible and investigators of the study 3- All participants will practice on the model first
  4-Responsible investigators will practice and show on the real patient.
  5-Then all participants will perform the application on the real patient under the supervision of responsible and investigators.
  Tracheal intubation time, success rate, number of interventions will be recorded by responsible and investigators.
  Interventions: Other: other

INTERVENTIONS:
Other: other — Our hypothesis is that playing video games may have positive effects on videostile use, but there is no research on this subject Our goal is to compare the performances of anesthesia assistants who have played video games with those who did not.

SUMMARY:
Video games are activities that require actively hand-eye coordination and where 3D thinking is at the forefront.

During the teaching of both laparoscopic surgery and robotic surgery techniques, it was revealed by the studies that the participants who played video games completed the trainings more easily and the success rate increased.

In a study comparing fiberoptic intubation success, anesthesia assistants playing video games had higher successful intubation rates and shorter intubation times in the first attempt.

Video stylets are newly developed devices that allow the use of video technology in airway management.

It has a camera at the end and a monitor to which the image is transferred. By transferring the real-time view of the airway structures, tracheal intubation increases the success rate and shortens the intubation time.

In order to determine whether video game playing has positive effects on videostylet use,ıt was aimed to compare the performances of the assistants who did play with the video game assistants.

DETAILED DESCRIPTION:
Anesthesiology assistants will be questioned about whether participants have played video games before or not.

Participants will be divided into two different groups as those with and without prior video game experience.

Video game will be played for those who have previous experience for 5 days via 0.5 hour mobile phone (Pubg mobile).No games will be played on the other group.

Then, all participants will be trained on the video stylet.

Within the scope of this training, all participants will watch videos about 1-Video stylet application.

2-Verbal explanation will be made by the responsible and investigators of the study 3- All participants will practice on the model first

4-Responsible investigators will practice and show on the real patient.

5-Then all participants will perform the application on the real patient under the supervision of responsible and investigators.

Tracheal intubation time, success rate, number of interventions will be recorded by responsible and investigators.

ELIGIBILITY:
Inclusion Criteria:

* Mallampati score I-II
* Cormack-Lehane score I-II
* ASA physical status I-II
* who required endotracheal intubation for elective surgery

Exclusion Criteria:

* Pregnancy
* Mallampati score III-IV
* Cormack-Lehane score III-IV
* ASA physical score III-IV
* sternomental distance < 12.5 cm
* mandibular-hyoid distance < 6 cm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo general anesthesia under elective conditions and have endotracheal intubation and who do not meet difficult intubation criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2020-06-25 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of video game playing habit in gaining videostyle-mediated intubation skill | 2 months
  tracheal intubation time

IPD SHARING:
Plan to Share IPD: No